CLINICAL TRIAL: NCT06670404
Title: PROTECT - Prospective Evaluation of Therapeutic Combination in Treating Vertebral Compression Fractures
Brief Title: Prospective Evaluation of Therapeutic Combination in Treating Vertebral Compression Fractures
Acronym: PROTECT
Status: Recruiting | Type: Observational
Sponsor: Prof Nicolas Theumann (Other)
Collaborators: Johnson & Johnson (Industry); Dr Danoob Dalili (Unknown)
Responsible Party: Sponsor-Investigator, Prof Nicolas Theumann, Professor, Hirslanden Clinique Bois-Cerf Lausanne
Organization: Hirslanden Clinique Bois-Cerf Lausanne (Other)
Other Study IDs: THU-2023-010
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Vertebral Compression Fractures; Pathological Fracture; Facet Joint Arthropathy
Keywords: vertebroplasty; CONFIDENCE High Viscosity Spinal Cement; observational post-market study
MeSH Terms: conditions — Fractures, Spontaneous | interventions — Vertebroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Vertebroplasty cohort: Patients with vertebral compression fractures treated with vertebroplasty
  Interventions: Device: Vertebroplasty

INTERVENTIONS:
Device: Vertebroplasty — Vertebral compression fractures treated with CONFIDENCE High Viscosity Cement

SUMMARY:
The purpose of this study is to collect clinical and radiographic outcomes in patients undergoing vertebroplasty procedures for the treatment of osteoporotic or pathological fractures of the vertebral body to understand the role of sagittal balance in patient outcomes. To support this objective, the sagittal balance measurement of sagittal vertical axis (SVA), NRS back pain, Quebec Back Pain Disability Scale (Quebec) score, and complications will be collected. The secondary purpose of the study is to review the role of sagittal balance and adjacent facet joint arthropathy treatment in patients with vertebral body fractures due to osteoporosis or tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years.
* Patients requiring vertebroplasty for the fixation of symptomatic pathological fractures of the thoracic or lumbar vertebral body resulting from osteoporosis or tumor.
* Symptomatic vertebral compression fracture(s) confirmed by MRI with bone marrow oedema on T2/STIR sequences.
* Diagnosis of osteoporosis (clinically and confirmed on DXA with quantifiable BMD) or pathological fracture due to tumor
* Patients with 1 or more vertebral compression fractures of the thoracic or lumbar spine Note: Patients with a current vertebral compression fracture who also have a previous history of vertebral compression fractures of the thoracic or lumbar spine may be included.

Study Specific Inclusion Criterion • Signed informed consent

Exclusion Criteria:

* Infection
* Vertebral body collapse to less than 1/3 (33%) of original height
* Vertebral plana (>90% vertebral body collapse)
* Spinal stenosis (retro pulsed fragments).
* Unstable spine warranting surgical stabilization
* Prophylactic treatment of any vertebrae with vertebroplasty
* Irreversible life threating bleeding disorders
* End stage kidney disease
* Drug dependence (IVDU)
* Pregnancy

Study Specific Exclusion Criterion:

• Unable or unwilling to follow the standard of care prescribed follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with vertebral compression fractures from osteoporosis or tumor eligible to be treated with vertebroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of sagittal balance | Up to 12 months post index surgery
  measurement of sagittal vertical axis (SVA)

SECONDARY OUTCOMES:
Improvement in Back Pain | Up to 12 months post index surgery
  Measured as NRS scale for back pain
Quebec Score | 6-12 months post index surgery
  Measured as the standard Quebec Score
Complications | Up to 12 months post-index surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Bois Cerf, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided